CLINICAL TRIAL: NCT02402452
Title: A Phase 1 Open-Label, Parallel-Group, Single-Dose Study to Evaluate the Pharmacokinetics of GS-9857 in Subjects With Normal Renal Function and Severe Renal Impairment
Brief Title: Pharmacokinetics of Voxilaprevir in Adults With Normal Renal Function and Severe Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-338-1125; 2015-000341-23 (EudraCT Number)
Record Dates: First submitted 2015-03-25; First posted 2015-03-30 (Estimated); Results first posted 2020-03-20 (Actual); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: HCV Infection
MeSH Terms: conditions — Hepatitis C | interventions — voxilaprevir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Renal Function (Experimental): Participants will receive a single dose of voxilaprevir on Day 1.
  Interventions: Drug: Voxilaprevir
- Severe Renal Impairment (Experimental): Participants will receive a single dose of voxilaprevir on Day 1.
  Interventions: Drug: Voxilaprevir

INTERVENTIONS:
Drug: Voxilaprevir — 100 mg tablet administered orally
  Other Names: GS-9857

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetics, safety, and tolerability of voxilaprevir (formerly GS-9857) in participants with severe renal impairment and matched healthy control participants.

ELIGIBILITY:
Key Inclusion Criteria:

* All individuals:

  * Screening laboratory values within defined thresholds for group
  * Use of two effective contraception methods if female of childbearing potential or sexually active male
* For individuals with severe renal impairment:

  * Stable chronic kidney disease
  * Creatinine clearance (CLcr) < 30 mL/min

Key Exclusion Criteria:

* All individuals:

  * Pregnant or nursing female or male with pregnant female partner
  * Hepatitis B virus, hepatitis C virus (HCV) or HIV infection
  * History of clinically significant illness or any other medical disorder that may interfere with the individual's treatment, assessment or compliance with the protocol
* For individuals with severe renal impairment:

  * Anticipated to require dialysis within 90 days of study dosing

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-05-05 (Actual); Primary Completion 2015-09-28 (Actual); Study Completion 2015-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, MD, PhD, Study Director — Gilead Sciences
Locations (4):
- United States (2):
  - Orlando Clinical Research Center, Orlando, Florida
  - Texas Liver Institute, San Antonio, Texas
- APEX GmbH, München, Germany
- Christchurch Clinical Studies Trust Ltd, Christchurch, New Zealand

REFERENCES:
- [Result] Lawitz E, Marbury T, Kirby BJ, Au NT, Mathias A, Stamm LM, Wei H, Sajwani K, Klein G, Gane E, Robson R. The effect of renal or hepatic impairment on the pharmacokinetics of GS-9857, a pangenotypic HCV NS3/4A protease inhibitor. The International Liver Congress; 2016; Barcelona, Spain.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States, Germany, and New Zealand. The first participant was screened on 05 May 2015. The last study visit occurred on 28 September 2015.
Pre-assignment Details: 39 participants were screened.
Groups:
- Severe Renal Impairment: Participants with severe renal impairment received a single dose of voxilaprevir 100 mg tablet orally on Day 1.
- Normal Renal Function: Participants with matched normal renal function received a single dose voxilaprevir of 100 mg tablet orally on Day 1.
Period: Overall Study
Arm/Group | Severe Renal Impairment | Normal Renal Function
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Severe Renal Impairment | Normal Renal Function | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Median (Standard Deviation); unit: years] | 59 (16.0) | 55 (14.1) | 57 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 8 | 8 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Black | 1 | 0 | 1
  Native Hawaiian or Pacific Islander | 0 | 0 | 0
  White | 9 | 10 | 19
  Not Permitted | 0 | 0 | 0
  Other | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 10 | 8 | 18
  Not Permitted | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 4 | 4 | 8
  New Zealand | 3 | 3 | 6
  United States | 3 | 3 | 6
Creatinine Clearance [Mean (Standard Deviation); unit: mL/min] | 21.2 (5.75) | 114.8 (15.31) | 68.0 (49.34)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.2 (5.54) | 26.6 (4.08) | 26.4 (4.74)

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter of Voxilaprevir: AUClast
Description: AUClast is defined as the area under the plasma concentration versus time curve from time zero to the last quantifiable concentration. Data presented are unadjusted geometric means and confidence intervals.
Time Frame: 0 (predose ≤ 5 min) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, 96, and 120 hours postdose
Population: PK Analysis Set included all enrolled participants who took at least 1 dose of study drug and had at least 1 nonmissing postdose concentration value reported by the PK laboratory for the corresponding analyte.
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Severe Renal Impairment | Normal Renal Function
Number analyzed (Participants) | 10 | 10
h*ng/mL | 662.7 [361.4 to 1215.3] | 383.3 [252.3 to 582.3]
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Normal Renal Function; An analysis of variance (ANOVA) appropriate for a parallel design was fitted to the natural logarithmic transformation of voxilaprevir AUClast. A 90% confidence interval (CI) was constructed for the geometric least squares mean (GLSM) ratio of AUClast for the comparison groups using two 1-sided tests; Test type: Other; Geometric Least-Square Mean(GLSM)Ratio % = 172.92, 90% CI 2-sided [97.93 to 305.33]

2. Primary Outcome: PK Parameter of Voxilaprevir: AUCinf
Description: AUCinf is defined as the area under the plasma concentration versus time curve extrapolated to infinite time. Data presented are unadjusted geometric means and confidence intervals.
Time Frame: 0 (pre-dose ≤ 5 minutes), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, 96, and 120 hours postdose
Population: Participants in the PK Analysis Set were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: h*ng/mL
Arm/Group | Severe Renal Impairment | Normal Renal Function
Number analyzed (Participants) | 10 | 10
h*ng/mL | 772.1 [426.3 to 1398.6] | 450.8 [295.7 to 687.4]
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Normal Renal Function; An ANOVA appropriate for parallel design was fitted to the natural logarithmic transformation of voxilaprevir AUCinf. A 90% CI was constructed for the GLSM ratio of AUCinf for the comparison groups using two 1-sided tests; Test type: Other; GLSM Ratio (%) = 171.27, 90% CI 2-sided [97.65 to 300.38]

3. Primary Outcome: PK Parameter of Voxilaprevir: Cmax
Description: Cmax is defined as the maximum observed plasma concentration of drug. Data presented are unadjusted geometric means and confidence intervals.
Time Frame: 0 (pre-dose ≤ 5 minutes), 0.25, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 24, 48, 72, 96, and 120 hours postdose
Population: Participants in the PK Analysis Set were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Severe Renal Impairment | Normal Renal Function
Number analyzed (Participants) | 10 | 10
ng/mL | 49.2 [26.6 to 91.1] | 33.9 [23.8 to 48.2]
Statistical Analysis 1: Comparison: Severe Renal Impairment vs Normal Renal Function; An ANOVA appropriate for parallel design was fitted to the natural logarithmic transformation of voxilaprevir Cmax. A 90% CI was constructed for the GLSM ratio of Cmax for the comparison groups using two 1-sided tests; Test type: Other; GLSM Ratio (%) = 145.43, 90% CI 2-sided [83.77 to 252.48]

4. Secondary Outcome: Percentage of Participants Who Experienced Treatment-Emergent Adverse Events (TEAE) and Laboratory Abnormalities
Description: The percentage of participants experiencing any TEAE or treatment-emergent laboratory abnormality was summarized.
Time Frame: First dose date to Day 31
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Severe Renal Impairment | Normal Renal Function
Number analyzed (Participants) | 10 | 10
percentage of participants
  Any TEAE | 20 | 50
  Any treatment-emergent laboratory abnormality | 70 | 30

ADVERSE EVENTS:
Time Frame: First dose date up to 31 days
Description: Safety Analysis Set included all participants who took at least 1 dose of study drug.
Arm/Group | Severe Renal Impairment | Normal Renal Function
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 2/10 | 5/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Severe Renal Impairment (N=10) | Normal Renal Function (N=10)
Constipation (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Vessel puncture site bruise (General disorders) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years